CLINICAL TRIAL: NCT04349683
Title: Efficacy and Safety of Jinshuibao for Patients With Chronic Kidney Disease Due to Glomerulonephritis：A Multicenter Randomized Controlled Clinical Trial
Brief Title: Efficacy and Safety of Jinshuibao for Patients With Chronic Kidney Disease Due to Glomerulonephritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jemincare (Industry)
Collaborators: Shanghai 6th People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NE-JSB-01
Record Dates: First submitted 2020-04-15; First posted 2020-04-16 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Chronic Kidney Disease Stage 3B; Chronic Kidney Disease stage4; Glomerulonephritis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Glomerulonephritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): basic treatment combined with Jinshuibao
  Interventions: Drug: Jinshuibao
- Control group (Placebo Comparator): basic treatment and placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Jinshuibao — 6 capsules at a time, 3 times a day (tid).
  Other Names: basic treatment
  Arms: Experimental group
Drug: Placebo — 6 capsules at a time, 3 times a day (tid).
  Other Names: basic treatment
  Arms: Control group

SUMMARY:
This is a multicenter, double-blind randomized controlled study to assess the efficacy and safety of Jinshuibao for patients with CKD due to glomerulonephritis, with a planned follow-up of 48 weeks.

DETAILED DESCRIPTION:
Previous studies have shown that cordyceps sinensis can act on several immune response pathways. Jinshuibao capsule, which is composed of fermented cordyceps sinensis powder (Cs-4) , has shown therapeutic effects in chronic kidney disease (CKD) according to small sample exploratory studies. Here, we conduct a prospective, double-blind randomized controlled study to assess the efficacy and safety of Jinshuibao for patients with CKD due to glomerulonephritis.

ELIGIBILITY:
Inclusion Criteria:

1. Aged >= 18 years old and <= 70 years old.
2. Patients with chronic kidney disease caused by primary glomerulonephritis diagnosed by previous pathology or diagnosed by clinician.
3. Chronic kidney disease stage 3b-4, that is, patients with eGFR between 15 and 45 ml/min per 1.73 m2 (according to 2012 KDIGO standard).
4. 24-hour urinary protein < 3g during the screening period.
5. Blood pressure, glucose, lipid and uric acid were measured during the screening period and were all in the following range: blood pressure: systolic blood pressure <140 and diastolic blood pressure < 90 mmHg; fasting blood-glucose < 8.0mmol/L or HbA1c < 8.0%; LDLl-c < 100 mg /dl (2.59 mmol/L), and TC < 230 mg /dl (5.95 mmol/L); uric acid < 420 mol/L.
6. Patients who have signed the informed consent.

Exclusion Criteria:

1. Pregnant or lactating women, or women of reproductive age who are unwilling to take reliable contraceptive measures.
2. Allergy to Jinshuibao.
3. Treatment with natural cordyceps sinensis, artificial cordyceps sinensis, traditional Chinese medicine or proprietary Chinese medicine with known renal impairment in recent 2 weeks.
4. Treatment with glucocorticoids, immunosuppressants or tripterygium wilfordii preparations in recent 3 months, or patients who have been confirmed to be treated with glucocorticoids, immunosuppressants or tripterygium wilfordii preparations in the following months.
5. History of gastrointestinal impairment or gastrointestinal diseases which may significantly affect the absorption of the experimental drugs, such as confirmed active ulcer (Forrest grade II or more severe impairment), inflammatory bowel disease, malabsorption syndrome, uncontrollable diarrhea or history of gastrointestinal surgery.
6. History of organ transplant, including kidney transplant.
7. History of severe diseases of the heart, brain, liver, hematopoietic system or other serious diseases affecting survival, such as malignant tumors, myocardial infarction, unstable angina, stroke or transient ischemic attack in recent 6 months.
8. Patients whose disease progresses too rapidly judged by the clinician.
9. Enrolled in other trials in recent 3 months.
10. Patients who are assessed by investigator as unsuitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2020-04-30 (Estimated); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Change of estimated glomerular filtration rate | Baseline to 48 weeks
  Estimated Glomerular Filtration Rate (eGFR) will be calculated according to Chronic Kidney Disease Epidemiology Collaboration (CKD EPI) creatinine equation

SECONDARY OUTCOMES:
Change of surem creatinine and 24-hour urine protein | Baseline to 12 weeks, 24 weeks, 36 weeks, 48 weeks
  Surem creatinine (Scr) will be tested by a central laboratory
Change of urinary protein/creatinine ratio (PCR) | Baseline to 12 weeks, 24 weeks, 36 weeks, 48 weeks
  Change from baseline in PCR
Change of hs-CRP | Baseline to 24 weeks, 48 weeks
  Change from baseline in hs-CRP
Change of TNF-α, IL-1β, and IL-6 | Baseline to 24 weeks and 48 weeks
  Change from baseline in TNF-α, IL-1β, and IL-6
Time to decline of 50% in eGFR or development of ESRD, and incidence of decline of 50% in eGFR or development of ESRD | 48 weeks
  End stage renal disease (ESRD）is defined by the need for long-term dialysis or renal transplantation, or eGFR<15ml/min
Patients' Quality of life | Baseline to 24 weeks and 48 weeks
  Patients' Quality of life will be accessed by KDQOL-36 (Chinese Version)
Number of rehospitalizations | 48 weeks
  Number of rehospitalizations during the follow-up period